CLINICAL TRIAL: NCT02893982
Title: A Phase I Therapeutic Dose Escalation Study Using Percutaneous Image-Guided Navigation for High Dose Rate Brachyablation of Primary Liver Lesions
Brief Title: High Dose Rate Brachyablation of Primary Liver Lesions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was closed due to poor accrual
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Michael Folkert, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102014-018; NCI-2017-02248 (Registry Identifier: National Cancer institute)
Record Dates: First submitted 2016-09-02; First posted 2016-09-09 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- brachytherapy (Experimental): image-guided navigation of catheter placement for high dose rate (HDR) brachytherapy treatment of patients with primary liver lesions
  Interventions: Radiation: brachytherapy

INTERVENTIONS:
Radiation: brachytherapy — image-guided navigation of catheter placement for high dose rate (HDR) brachytherapy treatment of patients with primary liver lesions

SUMMARY:
The objectives of this study are to demonstrate feasibility of an optimized, image-guided pre-planned workflow to deliver at least 25 Gy to the periphery of the target lesion while maintaining established dose constraints to normal tissues, and to determine the maximum tolerated dose (MTD) while evaluating treatment delivery, safety, and efficacy utilizing a pre-planned and optimized image-guided workflow for percutaneous HDR brachytherapy of liver lesions.

DETAILED DESCRIPTION:
Primary endpoints of this protocol are to demonstrate feasibility of an optimized, image-guided pre-planned workflow to deliver at least 25 Gy to the periphery of the target lesion while maintaining established dose constraints to normal tissues, and then to determine the maximum tolerated dose (MTD) of navigated percutaneous interstitial HDR brachytherapy for liver lesions. Secondary endpoints include assessment of toxicity and oncologic outcome (primarily local control at the treated site) and exploratory endpoints will be supported by advanced imaging studies at the time of the treatment procedure.

The 25 Gy starting dose was chosen as it has been shown to be effective at controlling tumor, albeit with limited followup. The promising outcomes noted at that dose are predicated on actually delivering that dose, hence the feasibility endpoint for meeting the goal dose delivery. While the other primary endpoint will be toxicity so as to avoid exceeding the MTD, this trial will treat more patients at each level to better characterize both toxicity and efficacy within a dose level (the therapeutic window). The investigators will attempt to escalate to levels that modeling would predict to have durable local control approaching 100%.55 Dose escalation levels of 5 Gy were chosen to mirror other studies performed at this institution with SBRT

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic or radiographic proof of a primary liver malignancy suitable for radiation therapy.
* Lesion size ≥ 3cm in maximum dimension.
* Predicted survival of >6 months.
* KPS ≥ 60 (See Appendix B).
* Age ≥ 18 years old.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.
* Formal evaluation by the Liver Tumor Program at UTSW: All patients should be fairly and prudently informed of their treatment options. To this end, all patients must be evaluated by the Liver Tumor Program at conference before brachytherapy treatment for discussion and consideration of other options for treatment of liver cancer including surgical resection.

Exclusion Criteria:

* Patients with a history of prior irradiation or other treatment to the liver or abdomen who after treatment on this protocol would have a cumulative dose to the liver or other normal tissues greater than the protocol defined constraints.
* Need or plans for concomitant antineoplastic therapy (including surgery, cryotherapy, radiofrequency ablation, chemo-embolization, conventionally fractionated radiotherapy, stereotactic body radiation therapy, and hepatic artery chemotherapy) for the protocol treated lesions except at progression. Adjuvant systemic therapy before and after the protocol therapy per section 4.4.1, and surgery or other ablative therapy is allowed for lesions appearing after enrollment to this protocol as per section 4.4.2 and 4.4.3 is allowed. At least 4 weeks must have passed since the last directed intervention to the protocol-treated lesion.
* Germ cell or hematologic malignancies.
* History of Crohn's Disease or Ulcerative Colitis.
* Active peptic ulcer disease for lesions within 5cm of the stomach.
* Underlying hepatic cirrhosis with Child-Pugh class B9 or C
* A major psychiatric illness which would limit understanding of the proposed protocol treatment and consent process.
* Men and women of reproductive potential may not participate unless they agree to use an effective contraceptive method.
* Pregnant or lactating women.
* Patients with parahepatic extension of disease with direct non-liver visceral involvement.
* Abnormal laboratory chemistries

  * Albumin < 2.5
  * Alkaline Phosphatase > 5 X upper limits of normal (ULN)
  * LT/AST > 5 X ULN
  * Total bilirubin > 5
* Abnormal complete blood count refractory to treatment. Any of the following:

  * Platelet count < 75,000/ml
  * Hb level < 8 gm/dl
  * ANC < 500/ml
* Abnormal coagulation profile: INR > 2 and/or PTT > 80

  * Patients who are on anticoagulation medication that may not be safely held for the procedure (≥ 5 days for antiplatelet agents and warfarin; ≥ 24 hours for low-molecular weight heparin formulations) will be excluded.
* Contraindications to general anesthesia
* Subjects receiving any other investigational agents.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
dosimetric coverage of liver lesions | 1 day
  Verify feasibility of HDR brachytherapy treatment and workflow for liver lesions using catheters placed under image-guided navigational techniques, to provide dosimetric coverage of liver lesions such that:
  1. Minimum CTV peripheral dose ≥ 25 Gy (D100 ≥ 25 Gy)
  2. 67% or 700 cc Liver < 5 Gy
  3. Esophagus, stomach, bowel, or duodenum < 15 Gy to 1cc, < 12 Gy to 5cc, < 9 Gy to 10cc, and 85 Gy in BED(2Gy) equivalent including current and prior treatment to 1cc
  4. Spinal cord/cauda equina < 8 Gy to 1 cc, or 75 Gy in 2 Gy fractions BED(2Gy) equivalent including current and prior treatment
  5. Kidney < 11 Gy, 200 cc < 8.4 Gy
  4. Spinal cord/cauda equina < 8 Gy to 1 cc, or 75 Gy in 2 Gy fractions BED(2Gy) equivalent including current and prior treatment 5. Kidney < 11 Gy, 200 cc < 8.4 Gy Verify feasibility of HDR brachytherapy treatment and workflow for liver lesions using catheters placed under image-guided navigational techniques
maximum tolerated dose | 90 days
  Determine the maximum tolerated dose (MTD) for percutaneous image-guided navigated high dose rate brachytherapy for liver lesions.
  1. Initial dose level; as above, minimum CTV peripheral dose ≥ 25 Gy
  2. Dose level 2: minimum CTV peripheral dose ≥ 30 Gy
  3. Dose level 3: minimum CTV peripheral dose ≥ 35 Gy

SECONDARY OUTCOMES:
severe toxicity | 30 days
  Demonstrate safety of HDR brachytherapy for lesions of the liver, defined as an acceptable level of severe toxicity (both acute and late effects) in the setting of HDR brachytherapy treatment. Severe toxicity will be defined as ≥ grade 3 Clavien-Dindo scale surgical complication score within 30 days of treatment or by NCI CTCAE v 4.0 toxicity after 30 days that is at least possibly related to treatment
local control | 2 years
  Assess patients for duration of local control at the treatment site, as well as other oncologic outcomes including progression-free and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Folkert, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No